CLINICAL TRIAL: NCT01009788
Title: A Phase 2 Study of ABT-888 and Temozolomide for Metastatic Breast Cancer and an Expansion Cohort in BRCA1/2 Mutation Carriers
Brief Title: ABT-888 and Temozolomide for Metastatic Breast Cancer and BRCA1/2 Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steven J Isakoff, MD, PhD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Steven J Isakoff, MD, PhD, Attending Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-261
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; BRCA1 Gene Mutation; brca2 Gene Mutation
Keywords: ABT-888; temozolomide; TMZ
MeSH Terms: conditions — Breast Neoplasms | interventions — veliparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TMZ/ABT888 Primary Cohort (Experimental): Primary cohort included patients unselected for BRCA1/2 mutations or breast cancer subtype.
  Combination therapy with temozolomide and veliparib (28 day cycle) Veliparib 30-40 mg orally twice/day days 1-7 Temozolomide 150 mg/m^2 orally once daily days 1-5, increased to 200 mg/m^2 starting cycle 2 as tolerated
  Interventions: Drug: ABT-888; Drug: temozolomide
- TMZ/ABT888 Expansion Cohort (Experimental): Expansion cohort included patients with BRCA1/2 deleterious mutations.
  Combination therapy with temozolomide and veliparib (28 day cycle) Veliparib 30 mg orally twice/day days 1-7 Temozolomide 150 mg/m^2 orally once daily days 1-5, increased to 200 mg/m^2 starting cycle 2 as tolerated
  Interventions: Drug: ABT-888; Drug: temozolomide

INTERVENTIONS:
Drug: ABT-888 — Capsules (30-40 mg) taken orally twice a day on days 1-7 of each 28 day cycle
  Other Names: veliparib
Drug: temozolomide — Capsules (150 mg/m^2 initially, and 200 mg/m^2 starting cycle 2 if tolerated) taken orally once a day on days 1 through 5 of a 28 day cycle
  Other Names: TMZ

SUMMARY:
The purpose of this research study is to find out if the combination of ABT-888 and temozolomide is safe and effective in treating patients with metastatic breast cancer. ABT-888 works by obstructing a DNA enzyme called poly (ADP-ribose) polymerase (PARP) which helps repair cancer cells damaged by chemotherapy. By blocking the PARP enzyme, the cancer cells are unable to repair themselves and as a result die. The other drug in this study is temozolomide. Temozolomide is designed to damage DNA in order to prevent cancer cells from reproducing. Because PARP inhibitors, such as ABT-888, prevent cancer cells from repairing their own DNA, they enhance the potential of chemotherapy therapy like temozolomide to induce cell death. The combination of ABT-888 and temozolomide has been used in a clinical trial for treatment of other cancers and information for this research study suggests that the combination may help to inhibit growth in breast cancer.

ONLY THE EXPANSION COHORT BELOW IS RECRUITING:

BRCA CARRIER EXPANSION COHORT: The purpose of the expansion cohort is to further evaluate the activity and safety of this combination in BRCA mutation carriers with metastatic breast cancer.

DETAILED DESCRIPTION:
* Each treatment cycle lasts 28 days. Participants will be given a supply of ABT-88 in the form of capsules which they will take twice daily on days 1-7 of each cycle. Temozolomide is also in capsule form and will be taken once daily on days 1-5 of each cycle.
* Participants will come into the clinic on day 1 of each cycle and will have the following tests and procedures performed: physical examination, vital signs and blood tests.
* On day 15 of cycles 1 and 2 and day 22 of each cycle, participants will have blood work done.
* An assessment fo the tumor by CT scan of the participants chest, abdomen and pelvis will be done every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer that is metastatic (Stage IV) or locally advanced recurrent breast cancer that is unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Measurable disease by RECIST criteria
* All immunohistochemical subtypes of breast cancer are eligible. HER2 positive breast cancer must have progressed on prior standard HER2 therapy or have a contraindication to anti-HER2 therapy.
* Must have at least 1 prior chemotherapy regimen for metastatic disease, with no limit on total number of prior therapies.
* 18 years of age or older
* Life expectancy of at least 12 weeks
* ECOG Performance Status of 0, 1, or 2
* Normal organ and marrow function as outlined in the protocol
* Archived tissue block or 25 unstained slides (from primary and/or metastatic tumor) if available for correlative exploratory studies. Absence of available tissue will not exclude the subjects from participating.
* CNS metastases are allowed if they are clinically stable without current evidence of symptomatic progression and do not require steroids, whole brain radiation therapy, or stereotactic radiosurgery. This may include brain metastases not previously treated if they are clinically stable as described above.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Women of child-bearing potential must have a negative pregnancy test within 14 days of registration.
* Patients must be progressing on their current therapy
* Prior exposure to single agent PARP inhibitor is allowed, but no prior exposure to PARP with a combination of chemotherapy is allowed.

Exclusion Criteria:

* Participants who have had chemotherapy, biologic therapy, small molecule targeted therapy or radiotherapy within 14 days prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. Anti-cancer hormonal therapy must be stopped 24 hours prior to starting study treatment.
* Participants may not be receiving any other investigational agents.
* Prior therapy with TMZ is allowed except if participant has a history of allergic reactions attributed to TMZ, or if therapy was discontinued due to intolerance of or toxicity from TMZ.
* Leptomeningeal disease
* CNS involvement requiring steroids (except for patients who recently completed brain radiation and are on stable or tapering doses of steroids).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, recent myocardial infarction, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, or other comorbid condition that investigator believes may compromise participant's safe and effective participation in the trial.
* Concurrent radiation therapy is not permitted while on study
* Concurrent anti-cancer therapy is not permitted on study
* Pregnant and breast feeding women
* History of uncontrolled seizure disorder
* Individuals with a history of other malignancies are eligible if they meet the following criteria: a) the other malignancy was treated with curative intent and is deemed by the investigator to be at low risk of recurrence , AND b) a metastatic lesion has been histologically confirmed as breast cancer, c) individuals with the following cancers are eligible if diagnosed and treated: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

EXPANSION COHORT:

An expansion cohort will have the same eligibility requirements with the following notable exceptions:

* Patients must have known deleterious mutation of BRCA1/2
* Prior PARP inhibitor combinations with chemotherapy are allowed
* Any number of prior therapies is allowed, including first line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Isakoff, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu J, Keenan TE, Overmoyer B, Tung NM, Gelman RS, Habin K, Garber JE, Ellisen LW, Winer EP, Goss PE, Yeap BY, Chabner BA, Isakoff SJ. Phase II trial of veliparib and temozolomide in metastatic breast cancer patients with and without BRCA1/2 mutations. Breast Cancer Res Treat. 2021 Oct;189(3):641-651. doi: 10.1007/s10549-021-06292-7. Epub 2021 Aug 20. PMID 34417675

RESULTS

PARTICIPANT FLOW:
Groups:
- TMZ/ABT888 Primary Cohort: Primary cohort included patients unselected for BRCA1/2 mutations or breast cancer subtype.
  Combination therapy with temozolomide and veliparib (28 day cycle) Veliparib 30-40 mg orally twice/day days 1-7 Temozolomide 150 mg/m^2 orally once daily days 1-5, increased to 200 mg/m^2 starting cycle 2 as tolerated
  ABT-888: Capsules (30-40 mg) taken orally twice a day on days 1-7 of each 28 day cycle
  temozolomide: Capsules (150 mg/m^2 initially, and 200 mg/m^2 starting cycle 2 if tolerated) taken orally once a day on days 1 through 5 of a 28 day cycle
- TMZ/ABT888 Expansion Cohort: Expansion cohort included patients with BRCA1/2 deleterious mutations.
  Combination therapy with temozolomide and veliparib (28 day cycle) Veliparib 30 mg orally twice/day days 1-7 Temozolomide 150 mg/m^2 orally once daily days 1-5, increased to 200 mg/m^2 starting cycle 2 as tolerated
  ABT-888: Capsules (30-40 mg) taken orally twice a day on days 1-7 of each 28 day cycle
  temozolomide: Capsules (150 mg/m^2 initially, and 200 mg/m^2 starting cycle 2 if tolerated) taken orally once a day on days 1 through 5 of a 28 day cycle
Period: Overall Study
Arm/Group | TMZ/ABT888 Primary Cohort | TMZ/ABT888 Expansion Cohort
Started | 42 | 21
Completed | 41 | 21
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMZ/ABT888 Primary Cohort | TMZ/ABT888 Expansion Cohort | Total
Number analyzed (Participants) | 41 | 21 | 62
Age, Continuous [Median (Full Range); unit: years] | 50 [31 to 68] | 46 [29 to 81] | 48 [29 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 21 | 61
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 35 | 18 | 53
  Unknown or Not Reported | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 31 | 16 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of ABT-888 and Temozolomide (TMZ) in Metastatic Breast Cancer
Description: Objective response rate (ORR) is defined as the percentage of enrolled patients who have a partial or complete response per RECIST (Response Evaluation Criteria in Solid Tumors) v1.1 guidelines. A partial response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. A complete response is defined as disappearance of all target lesions, with any pathological lymph nodes (whether target or non-target) reduced in short axis to <10 mm.
Time Frame: 2 years
Population: For the primary cohort, 7 patients were not evaluable out of the original 41 because they had no follow up imaging due to rapid clinical progression. For the expansion cohort, 3 patients were not evaluable out of the original 21 because they had no follow up imaging due to rapid clinical progression.
Measure: Count of Participants; unit: Participants
Arm/Group | TMZ/ABT888 Primary Cohort | TMZ/ABT888 Expansion Cohort
Number analyzed (Participants) | 34 | 18
Participants | 4 | 3

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the length of time from enrollment until disease progression, death, or date of last patient contact. Progressive disease was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progressive disease is defined as at least a 20% increase (at least 5 mm) in the sum of the LD of target lesions in comparison with the lowest sum achieved on study or the appearance of one or more new lesions, and/or unequivocal progression of non-target lesions.
Time Frame: 5 years
Measure: Median (Full Range); unit: months
Arm/Group | TMZ/ABT888 Primary Cohort | TMZ/ABT888 Expansion Cohort
Number analyzed (Participants) | 41 | 21
months | 1.8 [1.6 to 2.5] | 3.0 [2.1 to 6.2]

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) is defined as the percentage of patients who achieve a partial or complete response or stable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. A partial response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. A complete response is defined as disappearance of all target lesions, with any pathological lymph nodes (whether target or non-target) reduced in short axis to <10 mm. Progressive disease is defined as at least a 20% increase (at least 5 mm) in the sum of the LD of target lesions in comparison with the lowest sum achieved on study or the appearance of one or more new lesions, and/or unequivocal progression of non-target lesions.
Time Frame: Four months
Measure: Count of Participants; unit: Participants
Arm/Group | TMZ/ABT888 Primary Cohort | TMZ/ABT888 Expansion Cohort
Number analyzed (Participants) | 41 | 21
Participants | 11 | 9

ADVERSE EVENTS:
Time Frame: Up to 16 months
Arm/Group | TMZ/ABT888 Primary Cohort | TMZ/ABT888 Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 36/42 | 18/21
Serious Adverse Events (participants affected / at risk) | 25/42 | 4/21
Other Adverse Events (participants affected / at risk) | 42/42 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMZ/ABT888 Primary Cohort (N=42) | TMZ/ABT888 Expansion Cohort (N=21)
Increased alkaline phosphatase (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
arm pain (Musculoskeletal and connective tissue disorders) | 1 | 0
ascites (Gastrointestinal disorders) | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
bowel perforation (Gastrointestinal disorders) | 1 | 0
centralized abdominal pain (Gastrointestinal disorders) | 1 | 0
chest pain (General disorders) | 1 | 0
dehydration (Metabolism and nutrition disorders) | 1 | 0
disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
edema (General disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
GI Hemorrhage (Gastrointestinal disorders) | 0 | 1
Hematocrit (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
hypoxia (Reproductive system and breast disorders) | 2 | 0
Infection with unknown ANC, cerebrospinal fluid (Infections and infestations) | 0 | 1
Leak, cerebrospinal fluid (Nervous system disorders) | 0 | 1
left distal femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Left lower extremity weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
low platelet count (thrombocytopenia) (Blood and lymphatic system disorders) | 4 | 0
mood alteration/anxiety (Psychiatric disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
nocardia infection (Infections and infestations) | 1 | 0
pain (General disorders) | 2 | 0
Pericardial Effusions (malignant) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
pleural effusion (malignant) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
pneumonia (Infections and infestations) | 1 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pulmonary/upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rectal bleeding (Gastrointestinal disorders) | 1 | 0
Rectal proctitis (Gastrointestinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2
upper extremity pain right arm (Musculoskeletal and connective tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMZ/ABT888 Primary Cohort (N=42) | TMZ/ABT888 Expansion Cohort (N=21)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 42 | 20
Anxiety (Psychiatric disorders) | 1 | 2
Ascites (non-malignant) (Gastrointestinal disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 | 0
Blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 0 | 2
Blurred vision (Eye disorders) | 1 | 1
Coagulation disorders - other (Investigations) | 0 | 1
Constipation (Gastrointestinal disorders) | 41 | 20
Constitutional Symptoms - other (General disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Decreased Bone marrow cellularity (Blood and lymphatic system disorders) | 1 | 0
Decreased FEV (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decreased hemoglobin (Blood and lymphatic system disorders) | 41 | 20
Decreased leukocytes (Blood and lymphatic system disorders) | 41 | 20
Decreased neutrophils (Blood and lymphatic system disorders) | 40 | 21
Decreased platelets (Blood and lymphatic system disorders) | 42 | 20
decreased upper extremity function (Musculoskeletal and connective tissue disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 2
Depression (Psychiatric disorders) | 5 | 1
Dermatology/skin - other (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 41 | 20
Dizziness (Nervous system disorders) | 6 | 3
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Edema: limb (General disorders) | 3 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Eyelid dysfunction (Eye disorders) | 1 | 0
Fatigue (General disorders) | 42 | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 41 | 21
Fever (General disorders) | 41 | 21
Flu like syndrome (General disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal - other (Gastrointestinal disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Genitourinary obstruction (Renal and urinary disorders) | 1 | 0
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 41 | 20
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 | 1
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage, GI (lower GI NOS) (Gastrointestinal disorders) | 1 | 0
Hemorrhage, pulmonary/upper respiratory (Mediastinum) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hot flashes/flushes (Vascular disorders) | 0 | 2
Hyperbilirubinemia (Metabolism and nutrition disorders) | 5 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 14 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 41 | 20
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Hypertension (Vascular disorders) | 4 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 13 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 3
Hyponatremia (Metabolism and nutrition disorders) | 13 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 2
Hypotension (Vascular disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Increased alkaline phosphatase (Metabolism and nutrition disorders) | 19 | 5
Increased ALT (Metabolism and nutrition disorders) | 41 | 20
Increased AST (Metabolism and nutrition disorders) | 41 | 20
Increased creatinine (Investigations) | 2 | 0
Increased PTT (Partial Thromboplastin time) (Investigations) | 0 | 1
Infection - other (Infections and infestations) | 8 | 2
Insomnia (Psychiatric disorders) | 8 | 1
Joint-effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower extremity muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Lymphatics - other (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 15 | 4
Metabolic/laboratory - other (Metabolism and nutrition disorders) | 5 | 2
Mucositis (oral cavity) (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 42 | 21
Neurology - other (Nervous system disorders) | 1 | 0
Neuropathy: cranial (Nervous system disorders) | 2 | 0
Neuropathy: sensory (Nervous system disorders) | 8 | 0
Obstruction, GI (Ileum) (Gastrointestinal disorders) | 0 | 1
Ocular/visual - other (Eye disorders) | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (General disorders) | 41 | 20
Palpitations (Cardiac disorders) | 1 | 0
Perforation, GI (small bowel NOS) (Gastrointestinal disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1
Photophobia (Eye disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 41 | 20
Rash: Eythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 0
Speech impairment (Nervous system disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Sweating (diaphoresis) (General disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Upper extremity muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Voice changes (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 41 | 20
Watery eye (Eye disorders) | 1 | 0
Weight gain (General disorders) | 0 | 1
Weight loss (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-09-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT01009788/Prot_SAP_000.pdf